CLINICAL TRIAL: NCT02700789
Title: Pregnancies of Uncertain Location or Viability Research
Acronym: PULoVR
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 13008
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Intrauterine Pregnancy; Ectopic Pregnancy
Keywords: diagnostic accuracy; double decidual sac sign; intrauterine pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Women with a positive urinary pregnancy test following in vitro fertilisation/intracytoplasmic sperm injection (IVF/ICSI) treatment will be invited to attend for an additional transvaginal ultrasound scan at 33-34 days gestation. This will be conducted by a single investigator with experience in early pregnancy ultrasound using a Voluson E8 machine with a high frequency (5-9MHz and 9-12MHz) transvaginal probe and following standard operating procedures.
  Interventions: Procedure: Transvaginal ultrasound scan

INTERVENTIONS:
Procedure: Transvaginal ultrasound scan — The presence of the following structures will be recorded: an intrauterine fluid collection; the double decidual sac sign; yolk sac; and fetal pole.

SUMMARY:
Study to determine the diagnostic accuracy of the double decidual sac sign to predict an intrauterine pregnancy prior to ultrasonographic visualisation of embryonic contents using modern ultrasound technology.

DETAILED DESCRIPTION:
This diagnostic accuracy study will be conducted following the standards for reporting of diagnostic accuracy study (STARD) guidelines. Participants will be recruited from Nurture Fertility, Nottingham, United Kingdom at the time of embryo transfer. If the subsequent pregnancy test is positive, participants will be invited to attend for an additional transvaginal ultrasound scan at 33-34 days gestation. This scan will be considered to be the 'index test'.

The index test will be performed by a single investigator with experience in early pregnancy ultrasound following standard operating procedures using a Voluson E8 machine with a high frequency (5-9MHz and 9-12MHz) transvaginal probe. During the early scan the presence or absence of the following structures will be recorded: an intrauterine fluid collection (defined as a uniformly round, hypoechoic structure with an echogenic rim); the double decidual sac sign (DDSS) (defined as two concentric echogenic rings of tissue that surround the intraendometrial fluid collection that impress upon the endometrial stripe); yolk sac (defined as a spherical, hyperechoic ring situated eccentrically within the gestation sac); and fetal pole (defined as a small linear echogenic structure adjacent to the yolk sac, on the side closest to the gestational sac). If more than one intrauterine fluid collection is visualized then each will be considered as a separate entity. The findings from the early scan will be interpreted immediately and recorded separate to the main clinical notes. Participants will be excluded further from the study if at this point no intrauterine fluid collection is detected or if an intrauterine fluid collection containing a yolk sac or fetal pole is identified. Referral pathways to local Early Pregnancy Assessment Units (EPAU) will be in place for any woman in whom this early scan is strongly suggestive of an ectopic pregnancy, for example if there was an empty endometrial cavity and either an inhomogenous adnexal mass or an empty extra-uterine sac or a yolk sac or fetal pole with or without cardiac activity in an extra-uterine sac.

All women will then have a routine viability ultrasound scan at between 6 and 7 weeks gestation as per the fertility unit's standard practice. This viability scan was performed by an appropriately trained doctor or nurse following standard operating procedures and using the same ultrasound equipment as the index test. This viability scan plus any subsequent clinical follow-up required i.e. if the diagnosis was not certain following the viability scan alone, will constituted the reference standard. Clinical follow-up will consist of a repeat transvaginal ultrasound (TVS) 7-10 days after the initial viability scan in cases of pregnancies of uncertain viability (defined as the presence of an intrauterine gestation sac of less than 25mm mean diameter with no obvious yolk sac or fetal pole or an intrauterine gestation sac containing a fetal pole of less than 7mm with no obvious fetal heart pulsations) and in cases of pregnancies of uncertain location (defined as no evidence of an intra- or extra-uterine pregnancy or retained products of conception on transvaginal ultrasound scan in the presence of a positive urinary pregnancy test), referral to a local EPAU for monitoring of serial serum human chorionic gonadotropin (β-hCG) levels and subsequent ultrasonography and possibly surgery where indicated according to departmental protocols until a definitive diagnosis can be made. Interpretation of the reference standard will be performed by an experienced gynaecologist without knowledge of the findings from the index test. Any uncertainty regarding the final diagnosis will be dealt with by seeking the opinion of two other senior gynaecologists and gaining a consensus opinion.

The outcomes of interest are an intrauterine pregnancy (which may be viable or non-viable) or an ectopic pregnancy. A viable intrauterine pregnancy is defined as ultrasonographic identification of an intrauterine gestation sac with a fetal pole of any length with demonstrable fetal heart pulsations. A non-viable intrauterine pregnancy is defined as either an empty intrauterine gestation sac with mean sac diameter greater than 25mm or an intrauterine gestation sac containing a fetal pole with crown rump length greater than 7mm with no demonstrable fetal heart pulsations or in the absence of a viable embryo, no significant increase in the growth of the gestation sac or length of the fetal pole on two ultrasound scans performed more than 7 days apart. Where women undergo surgical or medical management of miscarriage, histological confirmation of the products of conception will be obtained when possible. Ectopic pregnancies will be confirmed either by direct visualisation during surgery with histological confirmation, or, in those managed medically with methotrexate or conservatively, unequivocal identification of an ectopic pregnancy on ultrasound scan. Ultrasonographic appearances indicative of an ectopic pregnancy will include: an empty endometrial cavity with either an inhomogenous adnexal mass or an empty extra-uterine sac or a yolk sac or fetal pole with or without cardiac activity in an extra-uterine sac. Following the reference standard, any pregnancy which does not fall into one of these categories will be excluded from the study. These included resolving or persisting pregnancies of unknown location.

The sensitivity and specificity of the DDSS for predicting an intrauterine pregnancy (IUP) will be estimated following cross tabulation of the index test results against those of the reference standard. The overall diagnostic accuracy, as well as positive and negative likelihood ratios and predictive values, will also be calculated. Results will be expressed as percentages for ease of interpretation and 95% confidence intervals will also be given.

ELIGIBILITY:
Inclusion Criteria:

* Positive urinary pregnancy test performed 18 days after oocyte retrieval in a fresh treatment cycle or 13-16 days after embryo transfer in a frozen embryo replacement cycle depending on the stage of embryo development at the time of transfer

Exclusion Criteria:

* Negative urinary pregnancy test performed 18 days after oocyte retrieval in a fresh treatment cycle or 13-16 days after embryo transfer in a frozen embryo replacement cycle depending on the stage of embryo development at the time of transfer
* No evidence of an intrauterine fluid collection during the index test
* Evidence of a yolk sac and/or fetal pole during the index test
* Final diagnosis not known

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited prospectively from Nurture Fertility, Nottingham, United Kingdom between 1st January and 31st October 2015. All women undergoing IVF/ICSI treatment will be invited to participate in the study.
  no ultrasonographic evidence of an intrauterine fluid collection, or a yolk sac and/or fetal pole was clearly visible within the intrauterine fluid collection. Women were also excluded if no outcome data were available or if, following the reference standard, the final diagnosis was not known (for example resolving or persistent pregnancies of unknown location).
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intrauterine Pregnancy | Repeat transvaginal ultrasound performed 8-16 days after the index test
  A viable intrauterine pregnancy is defined by ultrasonographic identification of an intrauterine gestation sac with a fetal pole of any length with demonstrable fetal heart pulsations. A non-viable intrauterine pregnancy is defined as either an empty intrauterine gestation sac with mean sac diameter greater than 25mm or an intrauterine gestation sac containing a fetal pole with crown rump length greater than 7mm with no demonstrable fetal heart pulsations or in the absence of a viable embryo, no significant increase in the growth of the gestation sac or length of the fetal pole on two ultrasound scans performed more than 7 days apart. Where women underwent surgical or medical management of miscarriage, histological confirmation of the products of conception will be obtained when possible.

SECONDARY OUTCOMES:
Ectopic Pregnancy | Repeat transvaginal ultrasound performed 8-16 days after the index test
  Ectopic pregnancies will be confirmed either by direct visualisation of an ectopic pregnancy during surgery with histological confirmation, or, in those managed medically with methotrexate or conservatively, unequivocal identification of an ectopic pregnancy on ultrasound scan. Ultrasonographic appearances indicative of an ectopic pregnancy include: an empty endometrial cavity with either an inhomogenous adnexal mass or an empty extra-uterine sac or a yolk sac or fetal pole with or without cardiac activity in an extra-uterine sac

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No